CLINICAL TRIAL: NCT07018310
Title: Micro Assays for HemATology Malignancies Antibody Treatment
Acronym: MAHATMAt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM25_0145; 2025-A01044-45 (Other: APHM)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood sampling (Experimental): blood sampling in patients with hematological malignancies
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Additional blood sampling as part of routine care

SUMMARY:
Hematological malignancy is a disease of the blood. In some cases, this pathology requires therapeutic management, which is not necessarily the case for you. Nevertheless, to improve the management of patients who need it, we are conducting research to assess the state of your immune system. Indeed, the role of the immune system is not limited to controlling infections, but is also important in controlling the proliferation of cancer cells, in hematology as in other types of cancer. Your immune system can play a spontaneous anti-tumor control role, but some so-called "immunotherapy" treatments aim to destroy cancer cells by stimulating the immune system, restoring its capabilities, and directing the immune response against tumor cells. For this immunotherapy treatment to be effective, since it uses your own immune cells (in most cases), these cells must be in a state to respond and be able to destroy the tumor. It is this ability to activate immune cells that is tested in this research protocol, using a simple test that could in future be used in routine clinical practice. But to understand why these immune cells don't work, we will also have to carry out genetic tests to analyze the various molecules that could interfere with the immune response, and try to inhibit the molecules that prevent the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years of age
* Patient with a hematological malignancy likely to benefit from immunotherapy (in any form; at the discretion of the referring physician)
* Before the start of 1st-line treatment, successive lines or before autograft (chemotherapy-free for at least 4 weeks in these cases).
* Patient has received information about the study and has not expressed opposition.
* Patient who is a beneficiary or entitled beneficiary of a social security scheme

Exclusion Criteria:

* Person in a period of exclusion from another research protocol at the time the non-opposition is signed.
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code, i.e. :

  * Persons deprived of their liberty by judicial or administrative decision
  * Persons subject to psychiatric monitoring under articles L3112-1 and L3113-1 who are not covered by the provisions of article L1121-8
  * Minors
  * Adults under legal protection or unable to express their consent.
* A person who cannot read and understand the French language well enough to be able to consent to take part in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Percentages of immune effectors | At the enrollement in the study
  Percentages of immune effectors responding to stimulation, assessed in patients with hematological malignancies

SECONDARY OUTCOMES:
Activation percentages (cytometry) vs. polymorphism expression percentage (molecular biology) | At the enrollement
  Analysis and comparison of activation percentages (cytometry) vs. polymorphism expression percentage (molecular biology)

CONTACTS AND LOCATIONS:
Locations (1):
- Assisitance Publique Hôpitaux de Marseille, Marseille, France